CLINICAL TRIAL: NCT02024464
Title: A Prospective, Multicenter, Randomized Comparison of the Hydrus Microstent to the iStent for Lowering Intraocular Pressure in Glaucoma Patients Undergoing Cataract Surgery
Brief Title: Comparing Hydrus Microstent(TM) to the iStent for Lowering IOP in Glaucoma Patients Undergoing Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivantis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-10-002
Record Dates: First submitted 2013-12-20; First posted 2013-12-31 (Estimated); Results first posted 2024-06-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliative Glaucoma; Pigmentary Dispersion Glaucoma
Keywords: Primary open angle glaucoma; POAG; Pseudoexfoliative glaucoma; PXG; Pigmentary dispersion glaucoma; PDG; Hydrus
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Lenses, Intraocular; Drug Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrus Microstent (Experimental): Cataract removal and intraocular lens (IOL) implantation, followed by insertion of the Hydrus Microstent in one eye (study eye)
  Interventions: Device: Hydrus Microstent; Procedure: Cataract removal and intraocular lens (IOL) implantation
- iStent (Active Comparator): Cataract removal and intraocular lens (IOL) implantation, followed by insertion of the iStent Trabecular Micro Bypass in one eye (study eye)
  Interventions: Device: iStent Trabecular Micro Bypass; Procedure: Cataract removal and intraocular lens (IOL) implantation

INTERVENTIONS:
Device: Hydrus Microstent — Device inserted into Schlemm's canal to enhance aqueous flow from the anterior chamber.
  Arms: Hydrus Microstent
Device: iStent Trabecular Micro Bypass — Device inserted into Schlemm's canal to enhance aqueous flow from the anterior chamber.
  Arms: iStent
Procedure: Cataract removal and intraocular lens (IOL) implantation — Cataract removal with phacoemulsification using standard techniques, followed by implantation with a posterior-chamber IOL suitable for glaucoma subjects

SUMMARY:
This clinical trial compares two implantable devices intended to lower the pressure inside the eye of glaucoma patients. One of the two devices will be implanted immediately following cataract surgery and the placement of a posterior chamber intra-ocular lens. Only one eye (study eye) will be implanted.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-masked, randomized clinical trial comparing Cataract Extraction (CE) + Hydrus Microstent to CE surgery + iStent implant for the reduction of intraocular pressure in patients with a positive diagnosis of primary open angle glaucoma, pseudoexfoliative glaucoma, or pigmentary dispersion glaucoma with an operable cataract. Eligible patients will be scheduled for cataract surgery. At the conclusion of successful cataract surgery and the placement of a posterior-chamber IOL, qualified subjects will be randomized to receive either the Hydrus Microstent or the iStent implant. Post-operative follow-up visits will be conducted at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary open angle glaucoma (POAG), Pseudoexfoliative (PXG) glaucoma, or Pigmentary dispersion glaucoma (PDG)
* An operable age-related cataract with BCVA of 20/40 or worse, eligible for phacoemulsification.

Exclusion Criteria:

* Forms of primary or secondary glaucoma not listed above
* Prior glaucoma surgery in the study eye

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-08; Primary Completion 2017-03 (Actual); Study Completion 2018-08 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and enrolled at 13 investigational sites outside of the United States
Pre-assignment Details: This reporting group includes all randomized patients (306).
Period: Overall Study
Arm/Group | Hydrus Microstent | iStent
Started | 154 | 152
Completed | 144 | 141
Not Completed | 10 | 11
Not completed — Discontinued | 5 | 4
Not completed — Missed Visits | 1 | 0
Not completed — Lost to Follow-up | 4 | 7

BASELINE CHARACTERISTICS:
Population: All randomized subjects, regardless of actual treatment received, procedure success, or compliance to protocol inclusion/exclusion criteria. [Intent-to-Treat (ITT)]
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrus Microstent | iStent | Total
Number analyzed (Participants) | 154 | 152 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.2) | 71.5 (7.5) | 72.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 71 | 157
  Male | 68 | 81 | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White European | 103 | 106 | 209
  Black or African Descent | 4 | 3 | 7
  Asian | 21 | 21 | 42
  Native North American | 1 | 0 | 1
  Hispanic/Latino/Central & South | 24 | 22 | 46
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Unmedicated Mean Diurnal Intraocular Pressure (DIOP) at Month 12
Description: Intraocular pressure (IOP) was measured using Goldmann applanation tonometry and averaged over the 8 am, 12 pm, and 4 pm time points. IOP was recorded in millimeters mercury (mmHg). The IOP assessment occurred after a protocol-specified wash-out period from all glaucoma medications.
Time Frame: Month 12: 8 am, 12 pm, 4 pm
Population: Intent-to-Treat (ITT) with verifiable data at visit. ITT subjects with secondary glaucoma or pressure lowering procedures, terminal wash-out exemptions, or missed diurnal IOP assessments are counted as failures for response metrics and are assigned a zero value for change in DIOP for the effectiveness endpoints.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent | iStent
Number analyzed (Participants) | 139 | 141
Number analyzed (eyes) | 139 | 141
mmHg | 16.9 (4.5) | 18.1 (4.9)

2. Secondary Outcome: Percentage of Subjects With 20% Reduction From Baseline in Unmedicated DIOP at Month 12
Description: as for outcome 1
Time Frame: Month 12: 8 am, 12 pm, and 4 pm
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent | iStent
Number analyzed (Participants) | 139 | 141
Number analyzed (eyes) | 139 | 141
percentage of subjects | 82.0 | 83.7

3. Secondary Outcome: Percentage of Subjects With Unmedicated DIOP of Not Less Than 5 mmHg and Not More Than 18 mmHg at Month 12
Description: as for outcome 1
Time Frame: Month 12: 8 am, 12 pm, 4 pm
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent | iStent
Number analyzed (Participants) | 139 | 141
Number analyzed (eyes) | 139 | 141
percentage of subjects | 68.3 | 67.4

4. Post Hoc Outcome: Percentage of Subjects With Unmedicated DIOP of Not Less Than 5 mmHg and Not More Than 18 mmHg at Month 24
Description: as for outcome 1
Time Frame: Month 24: 8 am, 12 pm, 4 pm
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent | iStent
Number analyzed (Participants) | 138 | 135
Number analyzed (eyes) | 138 | 135
percentage of subjects | 64.5 | 50.4

5. Post Hoc Outcome: Mean Change From Baseline in Unmedicated Mean Diurnal Intraocular Pressure (DIOP) at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12: 8 am, 12 pm, 4 pm
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent | iStent
Number analyzed (Participants) | 139 | 141
Number analyzed (eyes) | 139 | 141
mmHg | -8.7 (4.2) | -8.0 (4.1)

6. Post Hoc Outcome: Mean Change From Baseline in Unmedicated Mean Diurnal Intraocular Pressure (DIOP) at Month 24
Description: as for outcome 1
Time Frame: Baseline, Month 24: 8 am, 12 pm, 4 pm
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent | iStent
Number analyzed (Participants) | 138 | 135
Number analyzed (eyes) | 138 | 135
mmHg | -7.5 (4.5) | -6.9 (4.4)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of surgery to study exit, approximately 24 months. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: Adverse events as defined in this study protocol include all adverse events (AE) in the study eye. Only study eye adverse events were collected.
Groups:
- Hydrus Microstent: Cataract removal and intraocular lens (IOL) implantation, followed by insertion of the Hydrus Microstent in one eye (the study eye)
- iStent: Cataract removal and intraocular lens (IOL) implantation, followed by insertion of the iStent Trabecular Micro Bypass in one eye (the study eye)
Arm/Group | Hydrus Microstent | iStent
All-Cause Mortality (participants affected / at risk) | 4/154 | 3/152
Serious Adverse Events (participants affected / at risk) | 2/154 | 8/152
Other Adverse Events (participants affected / at risk) | 24/154 | 16/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrus Microstent (N=154) | iStent (N=152)
BCVA loss >/= 2 lines ETDRS >/= 3 months (Eye disorders) | 0 (0) | 1 (1) — Post-operative event. Study eye.
Epiretinal Membrane (Eye disorders) | 0 (0) | 1 (1) — Post-operative event. Study eye.
IOP Increase (Eye disorders) | 0 (0) | 1 (1) — Post-operative event. Study eye.
Uncontrolled Glaucoma (Eye disorders) | 2 (2) | 4 (4) — Post-operative event. Study eye.
Wet Age-Related Macular Degeneration (Eye disorders) | 0 (0) | 1 (1) — Post-operative event. Study eye.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrus Microstent (N=154) | iStent (N=152)
IOP Increase (Eye disorders) | 5 (5) | 10 (11) — Post-operative Event
Peripheral Anterior Synechia (Eye disorders) | 19 (19) | 6 (7) — Post-operative Event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that they shall not, without the Sponsor's prior written consent, independently publish, publicly disclose, present or discuss any results of or information pertaining to PI's activities conducted under this Agreement; unless the multi-center manuscript is not submitted for publication within one (1) year after completion of the trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02024464/Prot_SAP_000.pdf